CLINICAL TRIAL: NCT04319718
Title: A Randomized, Double Blinded Study of the Safety and Pharmacokinetics of Two Vaginal Film Formulations Containing the Integrase Inhibitor MK-2048
Brief Title: Safety and Pharmacokinetics of Two Vaginal Film Formulations Containing the Integrase Inhibitor MK-2048
Acronym: FAME103
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hillier, Sharon, PhD (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Katherine Bunge, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STUDY19100120; 1U19AI120249 (NIH)
Record Dates: First submitted 2020-03-17; First posted 2020-03-24 (Actual); Results first posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Pharmacokinetics; Safety
Keywords: Vagina; Film; Extended Release

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Eudragit MK-2048 vaginal film (Active Comparator): Single use of 2" x 2" vaginal film containing 30 mg of MK-2048 and 68.1 mg of ammonio methacrylate copolymer type B (Eudragit®).
  Interventions: Combination Product: MK-2048 High Eudragit Vaginal Film
- Low Eudragit MK-2048 vaginal film (Active Comparator): Single use of 2" x 2" vaginal film containing 30 mg of MK-2048 and 41.5 mg of ammonio methacrylate copolymer type B (Eudragit®).
  Interventions: Combination Product: MK-2048 Low Eudragit Vaginal Film

INTERVENTIONS:
Combination Product: MK-2048 High Eudragit Vaginal Film — 2" x 2" vaginal film containing 30 mg of MK-2048 and either 68.1 mg of ammonio methacrylate copolymer type B (Eudragit®)
  Arms: High Eudragit MK-2048 vaginal film
Combination Product: MK-2048 Low Eudragit Vaginal Film — 2" x 2" vaginal film containing 30 mg of MK-2048 and 41.5 mg of ammonio methacrylate copolymer type B (Eudragit®)
  Arms: Low Eudragit MK-2048 vaginal film

SUMMARY:
This is a proof of concept study to determine whether an extended release vaginal film can deliver drug for seven days. Two film formulations containing MK-2048 which differ by dissolution and spreadability attributes will be compared for safety and pharmacokinetic outcomes.

DETAILED DESCRIPTION:
This is a phase I randomized trial assessing the safety, acceptability, and pharmacokinetics of two formulations of MK-2048 vaginal film. While the primary objective is to evaluate the safety of the product, the overarching objective of this study is to provide proof of concept that an antiretroviral drug can be delivered in an extended release film formulation to provide drug delivery for 7 days or more after a single application. Forty eight women will be randomized with equal frequency to receive a single dose of a vaginal film containing MK-2048 (either the high Eudragit® or low Eudragit® formulation). The film will be inserted by a clinician on the day of enrollment. Vaginal swabs and plasma will be collected at days 0, 3, 5, 7, 10, 14 and 28 for all participants. On the day of enrollment, some participants may elect to participate in immediate post insertion sample collection (vaginal swab and plasma) at one or two time points within 6 hours of insertion. Genital biopsy samples and a rectal swab will be obtained on day 7, and cervicovaginal lavage will be collected at screening and days 14 and 28. The primary endpoint is the frequency of Grade 2 or higher adverse events. The secondary endpoints are: MK-2048 concentrations in plasma, cervical tissue homogenate, cervicovaginal lavage fluid, rectal and vaginal swab eluents; self-reported assessment of qualities of the experience with the films drawn from existing survey on microbicidal films, and general acceptability ratings drawn from market research methodology.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent.
* Willing to use an effective method of birth control throughout the duration of the study. Examples of effective methods include: hormonal methods (other than NuvaRing®), intrauterine device, bilateral tubal ligation, same sex partner, partner with a vasectomy, abstinence (defined as no vaginal sex for one month prior to screening).
* Able and willing to provide adequate locator information
* HIV-uninfected based on testing performed by study staff at screening
* In general good health as determined by the site clinician
* Agree to be sexually abstinent, including use of sex toys, from visit 2 (Enrollment) until visit 7 (7 days after the biopsy visit) and 48 hours prior to all study visits.
* Agree to refrain from use of vaginal device or products (for example, lubricants, creams, suppositories) throughout participation in the study. Tampons may be used except between visit 5 (biopsy visit) and visit 7 (day 14).
* Willingness to undergo all study-related assessments and follow all study-related procedures
* At screening and enrollment, agrees not to participate in other research studies involving drugs, medical devices, or vaginal products while enrolled in this trial
* Participants over the age of 21 (inclusive) must have documentation of a satisfactory Pap within three years prior to Enrollment consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 (Dated November 2007) to the Division of Acquired Immune Deficiency Syndrome Table for Grading Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017, or satisfactory evaluation with no treatment required of grade 1 or higher Pap results. If no documentation of a Pap smear can be provided, a Pap smear will be collected at the screening visit.

Exclusion Criteria:

* Menopause (as defined as amenorrhea for one year or more without an alternative etiology)
* Hysterectomy
* Participant report of any of the following:

  1. Known adverse reaction to any of the study products (ever)
  2. Non- therapeutic injection drug use in the 12 months prior to Screening
  3. Surgical procedure involving the pelvis in the 60 days prior to enrollment (includes dilation and curettage or evacuation, and cryosurgery; does not include cervical biopsy for evaluation of an abnormal pap smear)
  4. Participation in a drug, spermicide and/or microbicide study in the 30 days prior to enrollment
  5. Currently pregnant or pregnancy within 42 days prior to enrollment
  6. Currently lactating
  7. Use of a diaphragm, NuvaRing®, or spermicide for contraception
* Urogenital infection or suspected infection within 7 days of enrollment including: symptomatic candidiasis, trichomonas vaginalis, and symptomatic bacterial vaginosis; or cervical infection, including N. gonorrhoeae, C. trachomatis, or mucopurulent cervicitis; syphilis; herpes simplex virus lesions, or other sores (Note: seropositive herpes simplex virus without active lesions will not be excluded); acute pelvic inflammatory disease; urinary tract infection; recent exposure to a partner with N. gonorrhoeae, C. trachomatis, Trichomonas, syphilis, or non-gonorrheal urethritis
* Antibiotic or antifungal therapy (vaginal or systemic) within 7 days of enrollment
* As determined by the primary investigator, has any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine *including poorly controlled diabetes), respiratory, immunologic disorder or infectious disease
* Menses-like bleeding at the time of the Enrollment visit* or expected menses-like bleeding within 14 days of the Enrollment visit (*Women who have vaginal bleeding at the scheduled Enrollment visit may return at a different date to be re-examined and possibly enrolled provided they are still within the screening window and meet all criteria.)
* Any condition that, in the opinion of the Investigator, would preclude provision of consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Bunge, MD, Principal Investigator — University of Pittsburgh; Sharon L Hillier, PhD, Study Chair — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- High Eudragit MK-2048 Vaginal Film: Single use of 2" x 2" vaginal film containing 30 mg of MK-2048 and 68.1 mg of ammonio methacrylate copolymer type B (Eudragit®).
  MK-2048 High Eudragit Vaginal Film: 2" x 2" vaginal film containing 30 mg of MK-2048 and 68.1 mg of ammonio methacrylate copolymer type B (Eudragit®)
Period: Overall Study
Arm/Group | High Eudragit MK-2048 Vaginal Film | Low Eudragit MK-2048 Vaginal Film
Started | 25 | 12
Completed | 24 | 10
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Cervical biopsy not performed since participant did not refrain from sexual activity | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Eudragit MK-2048 Vaginal Film | Low Eudragit MK-2048 Vaginal Film | Total
Number analyzed (Participants) | 25 | 12 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (6.9) | 28.2 (5.5) | 27.2 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 12 | 37
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic, white | 2 | 0 | 2
  Non-Hispanic, white | 15 | 8 | 23
  Non-Hispanic, black | 3 | 1 | 4
  Asian | 2 | 1 | 3
  Bi-/multi-racial | 2 | 1 | 3
  Hispanic, not otherwise specified | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 25 | 12 | 37
Has current sexual partner [Count of Participants; unit: Participants] | 16 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 2 or Higher Adverse Events
Description: Number of participants who experience Grade 2 or higher adverse events
Time Frame: Through study completion, approximately 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Eudragit MK-2048 Vaginal Film | Low Eudragit MK-2048 Vaginal Film
Number analyzed (Participants) | 25 | 12
Participants | 2 | 5
Statistical Analysis 1: Comparison: High Eudragit MK-2048 Vaginal Film vs Low Eudragit MK-2048 Vaginal Film; Test type: Other; p = .025, Fisher Exact

2. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve of MK-2048
Description: Area under the plasma concentration versus time curve of MK-2048 reported as pg x day/mL. MK-2048 plasma concentration was measured at 0, 3, 5, 7, 10, 14, and 28 days after film insertion.
Time Frame: Through study completion, approximately 28 days
Measure: Median (Inter-Quartile Range); unit: pg x day/mL
Arm/Group | High Eudragit MK-2048 Vaginal Film | Low Eudragit MK-2048 Vaginal Film
Number analyzed (Participants) | 25 | 12
pg x day/mL | 1370 [706 to 2435] | 1873 [563 to 3959]
Statistical Analysis 1: Comparison: High Eudragit MK-2048 Vaginal Film vs Low Eudragit MK-2048 Vaginal Film; Test type: Other; p = .47, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Area Under the Cervical Tissue Homogenate Concentration Versus Time Curve of MK-2048
Description: Area under the cervical tissue homogenate concentration versus time curve of MK-2048 reported as pg x day/mL. MK-2048 concentration was measured at 0, 3, 5, 7, 10, 14, and 28 days after film insertion.
Time Frame: Through study completion, approximately 28 days
Population: MK 2048 levels in all tissue homogenate samples were below the limit of quantitation for the assay. Therefore, the area under the curve could not be calculated.
Measure: Median (Inter-Quartile Range); unit: pg x day/mL
Arm/Group | High Eudragit MK-2048 Vaginal Film | Low Eudragit MK-2048 Vaginal Film
Number analyzed (Participants) | 25 | 12
pg x day/mL | NA [NA to NA] — MK 2048 levels in all tissue homogenate samples were below the limit of quantitation for the assay. | NA [NA to NA] — MK 2048 levels in all tissue homogenate samples were below the limit of quantitation for the assay.

4. Secondary Outcome: Area Under the Cervicovaginal Lavage Fluid Concentration Versus Time Curve of MK-2048
Description: Area under the cervicovaginal lavage fluid concentration versus time curve of MK-2048 reported as pg x day/mL
Time Frame: Through study completion, approximately 28 days
Population: Data not collected
Arm/Group | High Eudragit MK-2048 Vaginal Film | Low Eudragit MK-2048 Vaginal Film
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Area Under the Rectal Swab Eluent Concentration Versus Time Curve of MK-2048
Description: Area under the rectal swab eluent concentration versus time curve of MK-2048 reported as pg x day/mL
Time Frame: Through study completion, approximately 28 days
Population: Data not collected
Arm/Group | High Eudragit MK-2048 Vaginal Film | Low Eudragit MK-2048 Vaginal Film
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Area Under the Vaginal Swab Eluent Concentration Versus Time Curve of MK-2048
Description: Area under the vaginal swab eluent concentration versus time curve of MK-2048 reported as ng x day/mL. MK-2048 concentration was measured at 0, 3, 5, 7, 10, 14, and 28 days after film insertion.
Time Frame: Through study completion, approximately 28 days
Measure: Median (Inter-Quartile Range); unit: ng x day/mL
Arm/Group | High Eudragit MK-2048 Vaginal Film | Low Eudragit MK-2048 Vaginal Film
Number analyzed (Participants) | 25 | 12
ng x day/mL | 543608 [50535 to 3256911] | 1112355 [58319 to 1642201]
Statistical Analysis 1: Comparison: High Eudragit MK-2048 Vaginal Film vs Low Eudragit MK-2048 Vaginal Film; Test type: Other; p = .67, Wilcoxon (Mann-Whitney)

7. Other Pre Specified Outcome: Median Fold Change in Percent Inhibition of Human Immunodeficiency Virus-1 Replication in Cervicovaginal Lavage Fluid
Description: Median fold change in in-vitro anti-human immunodeficiency virus-1 activity in cervicovaginal lavage fluid determined by the TZM-bl assay and defined as percent inhibition of human immunodeficiency virus-1 infection by luciferase for a single round of replication measured at day 28 divided by percent inhibition measured at baseline.
Time Frame: Through study completion, approximately 28 days
Population: All participants with a cervical biopsy sample taken. Two participants in the low Eudragit arm did not have cervical biopsies performed due to product discontinuation. One participant in the high arm also did not have a cervical biopsy collected due to safety concerns since she did not refrain from sexual activity prior to the visit.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | High Eudragit MK-2048 Vaginal Film | Low Eudragit MK-2048 Vaginal Film
Number analyzed (Participants) | 24 | 10
ratio | 1.01 [.13 to 1.25] | .92 [.09 to 1.11]
Statistical Analysis 1: Comparison: High Eudragit MK-2048 Vaginal Film vs Low Eudragit MK-2048 Vaginal Film; Test type: Other; p = .51, Wilcoxon (Mann-Whitney)

8. Other Pre Specified Outcome: Human Immunodeficiency Virus-1 p24 Core Protein Titer in Cervical Biopsies
Description: Human Immunodeficiency Virus-1 infection of cervical biopsies as defined as titer of the HIV-1 p24 core protein measured by ELISA and expressed as log10 pg/mL per mg of tissue
Time Frame: Through study completion, approximately 28 days
Population: All participants with a cervical biopsy sample taken. Two participants in the low Eudragit arm did not have cervical biopsies performed due to product discontinuation. One participant in the high Eudragit arm did not have a cervical biopsy collected due to safety concerns since she did not remain sexually abstinence prior to the visit and one participant's biopsy p24 results are not evaluable due to a lab processing error.
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | High Eudragit MK-2048 Vaginal Film | Low Eudragit MK-2048 Vaginal Film
Number analyzed (Participants) | 23 | 10
log10 pg/mL | 96.0 [17.1 to 1210.5] | 543.5 [265.0 to 9050.2]
Statistical Analysis 1: Comparison: High Eudragit MK-2048 Vaginal Film vs Low Eudragit MK-2048 Vaginal Film; Test type: Other; p = .09, Wilcoxon (Mann-Whitney)

9. Other Pre Specified Outcome: Mean Change in Nugent Score
Description: Mean change in the Nugent score as determined from vaginal smears. Nugent scores range from 0 to 10; 0 indicates a Lactobacillus-dominant microbiome while a score of 10 indicates a microbiome dominated by bacterial vaginosis-associated bacteria. Nugent scores were assessed at 0, 3, 5, 7, 10, 14, and 28 days after film insertion. The mean change was estimated from a mixed effects linear regression model and is defined as the average change between each post-insertion time point and the pre-insertion time point.
Time Frame: Through study completion, approximately 28 days
Population: All participants who had Nugent scores assessed at enrollment and at one or more follow-up visits. The 2 women who discontinued product in the low Eudragit arm were only followed for safety and did not have urogenital samples collected beyond the enrollment visit.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | High Eudragit MK-2048 Vaginal Film | Low Eudragit MK-2048 Vaginal Film
Number analyzed (Participants) | 25 | 10
units on a scale | -0.35 [-0.93 to 0.24] | -0.62 [-1.71 to 0.48]
Statistical Analysis 1: Comparison: High Eudragit MK-2048 Vaginal Film vs Low Eudragit MK-2048 Vaginal Film; Test type: Other; p = .65, Mixed Models Analysis
Statistical Analysis 2: Comparison: High Eudragit MK-2048 Vaginal Film; Test type: Other; p = .24, Mixed Models Analysis
Statistical Analysis 3: Comparison: Low Eudragit MK-2048 Vaginal Film; Test type: Other; p = .27, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | High Eudragit MK-2048 Vaginal Film | Low Eudragit MK-2048 Vaginal Film
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/12
Other Adverse Events (participants affected / at risk) | 17/25 | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Eudragit MK-2048 Vaginal Film (N=25) | Low Eudragit MK-2048 Vaginal Film (N=12)
Abnormal vaginal discharge (Reproductive system and breast disorders) | 8 (8) | 5 (5)
Vulvovaginal itching (Reproductive system and breast disorders) | 5 (5) | 4 (4)
Unexpected vaginal bleeding (Reproductive system and breast disorders) | 3 (3) | 4 (4)
Vulvovaginal irritation (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 2 (2)
Vaginal odor (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Early menses (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Back pain, low (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Post-traumatic stress disorder, worsening (Psychiatric disorders) | 0 (0) | 1 (1) — Post-traumatic stress disorder, worsening of pre-existing condition

LIMITATIONS AND CAVEATS:
After 25 participants were enrolled, 2 of 12 participants randomized to the low Eudragit® film arm had product discontinuations due to vaginal irritation and lack of product tolerability. The Protocol Safety Review Team voted to discontinue the low Eudragit® film arm resulting in only 12 participants of the 25 planned enrolled into that study arm. This limited the power of the study to detect significant differences in the outcomes between the two film arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT04319718/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT04319718/ICF_000.pdf